CLINICAL TRIAL: NCT03334370
Title: Evaluation of Quality of Care - Shared-Care Programme, HA
Acronym: QoC SCP
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Professor Cindy L.K. Lam, Clinical Professor, The University of Hong Kong
Other Study IDs: HKCTR-1185
Record Dates: First submitted 2017-10-24; First posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DM subjects in Hong Kong

SUMMARY:
Diabetes mellitus (DM) and hypertension (HT) are major causes of morbidity and among the top 10 causes of deaths in Hong Kong in 2008 (Department of Health 2009). The Hospital Authority (HA) has initiated service improvement through introducing the shared-care (SC) programme to improve the quality of care (QOC) for DM and HT patients. The evaluation on the QOC is an essential part of the programme in order to inform future policy. The Family Medicine Unit (FMU) of the University of Hong Kong (HKU) has been appointed by the HA to carry out the evaluation of the QOC of the programme.

The Action Learning and Audit Spiral methodologies to measure whether the target standard of care intended by the SC programme is achieved. Each SC participating clinic and private medical practitioner (PMP) will be invited to complete a structured evaluation questionnaire. The data of all patients who have enrolled into the programme will be included in the evaluation on the process and outcomes of care. A hundred and thirty participants will be followed up by telephone to evaluate the effect of the programme in quality of life (QOL), patient enablement, and global rating of change in health condition at baseline and 6 months after enrolment. Data on the process of care will be retrieved from the HA medical records.

Main Outcome Measures: The primary outcomes are the proportion of participants who received the criterion process of care and achieved a HbA1c level <7.5%.

Data Analysis: Descriptive statistics on proportions of clinics or subjects meeting the quality of care criteria will be calculated. The outcomes of SC patients will be compared at 6, 12, 24, 36 and 48 months by paired sample t-test. The outcomes between SC patients and control group will be compared by independent sample t-test or Chi-square test.

Hypothesis: The QOC of the SC programme will be determined. Areas of deficiency and possible areas for quality enhancement will be identified. The results of this study will provide empirical evidence on whether the HA's SC programme can achieve equivalent QOC as the usual HA care for diabetes mellitus (DM) patients. The information will be used to guide service planning and policy decision making.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes mellitus who have received care at the specialist outpatient clinic (SOPC)for at least 2 years, stratified to be of low risk and have normal renal function as defined by the plasma creatinine level.

Exclusion Criteria:

* Patients will be excluded if they are stratified to be at high cardiovascular risk or are suffering end stage renal failure, on dialysis or after transplantation, or on insulin, or do not give consent to be transferred.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetes mellitus who have received care at the specialist outpatient clinic (SOPC) for at least 2 years, stratified to be of low risk and have normal renal function as defined by the plasma creatinine level would be offered the option of being followed up by a private medical practitioner (PMP) in primary care with a financial subsidy and continuing support from the original SOPC. Each patient in the SC programme will receive an annual assessment and complication screening at the SOPC. The programme encourages long-term patient-doctor relationships in order to develop continuous and holistic care for CD patients. Patients will be excluded if they are stratified to be at high cardiovascular risk or are suffering end stage renal failure, on dialysis or after transplantation, or on insulin, or do not give consent to be transferred.
Sampling Method: Probability Sample
Enrollment: 620 (Actual)
Dates: Start 2010-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change of the proportion of clinics that have satisfied each of the structure criteria. | December, 2010; December, 2011; December, 2012; December, 2013; December, 2014
Change of the proportion of patients who have received with the SC criterion process of care. | June, 2011; December, 2011; December, 2012; December, 2013; December, 2014
Change of the proportion of patients who have achieved a HbA1c <7.5%. | June, 2011; December, 2011; December, 2012; December, 2013; December, 2014

SECONDARY OUTCOMES:
Low-density lipoprotein (LDL) | Baseline, 6, 12, 24, 36 and 48 months after enrollment.
Blood pressure (BP) | Baseline, 6, 12, 24, 36 and 48 months after enrollment.
Body mass index (BMI) | Baseline, 6, 12, 24, 36 and 48 months after enrollment.
Cardiovascular complications | Baseline, 6, 12, 24, 36 and 48 months after enrollment.
Patient reported outcomes (PRO) measured by the change in Short Form-12 version 2 (SF-12v2) scores at 6 months. | Baseline and 6 months after the first administration of questionnaire.
Patient reported outcomes (PRO) measured by the change in the Patient Enablement Instrument (PEI) scores at 6 months. | Baseline and 6 months after the first administration of questionnaire.
Patient reported outcomes (PRO) measured by the change in the Global Rating Scale (GRS) at 6 months. | Baseline and 6 months after the first administration of questionnaire.
Service utilization outcomes measured by General Outpatient Clinics (GOPC) attendance rates at baseline and 12, 24, 36 and 48 months after enrollment. | Baseline, 12, 24, 36 and 48 months after enrollment
Service utilization outcomes measured by specialist outpatient clinic (SOPC) attendance rates at baseline and 12, 24, 36 and 48 months after enrollment. | Baseline, 12, 24, 36 and 48 months after enrollment
Service utilization outcomes measured by accident & emergency (A&E) attendance rates at baseline and 12, 24, 36 and 48 months after enrollment. | Baseline, 12, 24, 36 and 48 months after enrollment
Service utilization outcomes measured by hospital attendance rates at baseline and 12, 24, 36 and 48 months after enrollment. | Baseline, 12, 24, 36 and 48 months after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hksar, Hong Kong